CLINICAL TRIAL: NCT07140211
Title: Short-term Low-dose Low-molecular-weight Heparin to Prevent Postpartum Thrombosis: a Pragmatic, Multi-center, Open-label Randomized Controlled Study
Brief Title: Short-term Low-dose Low-molecular-weight Heparin to Prevent Postpartum Thrombosis
Acronym: SHINE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Marc Blondon (Other)
Responsible Party: Sponsor-Investigator, Marc Blondon, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-00622
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Venous Thromboembolism (VTE); Postpartum
MeSH Terms: conditions — Venous Thromboembolism | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-molecular-weight heparin (Experimental)
  Interventions: Drug: Low-dose low-molecular-weight heparin
- No treatment (No Intervention)

INTERVENTIONS:
Drug: Low-dose low-molecular-weight heparin — Low-molecular-weight heparin given for 7-10 days after delivery:
  * enoxaparin 4000-6000IU o.d.
  * nadroparin 3800-5700IU o.d.
  * dalteparin 5000-7500IU o.d.
  * tinzaparin 4500-7000IU o.d.
  Arms: Low-molecular-weight heparin

SUMMARY:
The goal of this clinical trial is to evaluate the risk-benefit of a short-term treatment with a low-dose low-molecular-weight heparin (LMWH), in the postpartum period (after delivery). The main questions it aims to answer are:

* compared to no treatment, does short-term postpartum LMWH modify the risk of venous thromboembolism within 90 days of delivery?
* compared to no treatment, does short-term postpartum LMWH modify the risks of bleeding and wound complications? Participants will take low-dose LMWH for 7-10 days or no treatment, and will be followed for 90 days post-delivery.

ELIGIBILITY:
Inclusion Criteria: postpartum women after delivery AND ≥1 major risk factor / ≥2 minor risk factors:

* Major risk factors: Emergency cesarean section ; Pre-pregnancy BMI ≥35kg/m2 ; Known low-risk thrombophilia (heterozygous factor V Leiden; heterozygous G20210 prothrombin mutation) ; Pre-eclampsia ; Pre-term delivery ; Peripartum systemic infection ; Intra-uterine growth restriction ; Pregnancy loss
* Minor risk factors: Age ≥35 years ; Pre-pregnancy BMI 30.0-34.9kg/m2 ; Current smoking ; Elective cesarean section ; Postpartum hemorrhage ; Antenatal immobility

Exclusion Criteria:

* ≥2 doses of postpartum LMWH
* Any indication for therapeutic anticoagulation
* A high-risk of postpartum VTE
* An increased bleeding risk
* A contra-indication to heparin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Venous thrombotic outcomes | Within 90 days post-randomization
  Centrally-adjudicated, objectively-diagnosed, symptomatic venous thromboembolism (deep vein thrombosis / pulmonary embolism)

SECONDARY OUTCOMES:
All-cause mortality | Within 90 days post-randomization
Bleeding | Within 90 days post-randomization
  Obstetrical and non-obstetrical major and clinically-relevant non-major bleeding
Heparin-induced thrombocytopenia | Within 90 days post-randomization
Surgical site / perineal complications, and endometritis | Within 90 days post-randomization
Septic pelvic thrombosis | Within 90 days post-randomization
Superficial vein thrombosis | Within 90 days post-randomization
Stroke and cerebral vein thrombosis | Within 90 days post-randomization
Persistent lochia | At 42 day post-randomization
Maternal quality of life | At 14 days post-randomization
  Measured by the PROMIS global short form (PROMIS-10) questionnaire
Maternity clot risk | Within 90 days post-randomization
VTE surveillance (imaging) | Within 90 days post-randomization
Duration of hospital stay | Within 90 days post-randomization
Serious adverse events | Within 90 days post-randomization

OTHER OUTCOMES:
Main safety composite outcome | Within 90 days post-randomization
  Composite outcome of centrally-adjudicated obstetrical major bleeding, non-obstetrical major bleeding and/or major surgical site / perineal wound complication

IPD SHARING:
Plan to Share IPD: Undecided